CLINICAL TRIAL: NCT02108379
Title: An Open-label Outpatient In-season Study Assessing Compliance and Usability of Rhinix™ Nasal Filters
Brief Title: Compliance and Usability Study Evaluating RHINIX™ Nasal Filters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Rhinix ApS (Unknown); Astma-Allergi Danmark (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00002
Record Dates: First submitted 2014-03-18; First posted 2014-04-09 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-03

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rhinix Nasal Filters (Experimental): All included will receive rhinix nasal filters
  Interventions: Device: Rhinix Nasal Filters

INTERVENTIONS:
Device: Rhinix Nasal Filters

SUMMARY:
This study will investigate usability and compliance related to rhinix nasal filters for the treatment of seasonal allergic rhinitis (hay fever) during the natural grass pollen season in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Motivated to try a different treatment approach to seasonal allergic rhinitis (documented by answering the call-out by Astma-Allergi Danmark)
* Indicates having seasonal allergic rhinitis to grass via online questionnaire
* Informed consent (by email acceptance after having received information on the trial)
* Assess to internet and email

Exclusion Criteria:

* Improper fit of the Rhinix™ device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1073 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Week 1 likelihood of continued use of RHINIX after study end. | 1 assessment at the end of the 1st week of use.
  In week 1: The proportion of subjects that rate that they will definitely or are likely to continue using RHINIX after the study is over given that they have stated that they have tried the device.
Week 2 likelihood of continued use of RHINIX after study end. | 1 assessment at the end of the 2nd week of use.
  In week 2: The proportion of subjects that rate that they will definitely or are likely to continue using RHINIX after the study is over given that they have stated that they have tried the device.

SECONDARY OUTCOMES:
Week 1 Satisfaction with RHINIX | 1 assessment at the end of the 1st week
  In week 1: The proportion of subjects who are completely or somewhat satisfied with RHINIX given that they have used the product.
Week 2 satisfaction with RHINIX | One assessment at the end of the 2nd week
  In week 2: The proportion of subjects who are completely or somewhat satisfied with RHINIX given that they have used the product.
Week 1: RHINIX Control | One assessment at the end of the 1st week of use
  In week 1: The proportion of subjects who state that RHINIX has helped "to a very high degree" or "to a high degree" in controlling their hay fever symptoms given that they have used the product
Week 2: RHINIX Control | One assessment at the end of the 2nd week of use.
  In week 2: The proportion of subjects who state that RHINIX has helped "to a very high degree" or "to a high degree" in controlling their hay fever symptoms given that they have used the product

OTHER OUTCOMES:
Week 1: Correlation of use and allergy severiy | One assessment at the end of the 1st week of use
  In week 1: To assess the correlation between symptom severity at screening and likelihood of answering that they will definitely/likely continue using the product.
Week 2: Correlation between use and allergy severity | One assessment at the end of the 2nd week of use
  Week 2: To assess the correlation between symptom severity at screening and likelihood of answering that they will definitely/likely continue using the product.
Week 1: Perceived decrease in medication | One assessment after the 1st week of use
  In week 1: To assess whether use of RHINIX has led to a perceived decrease in use of medication.
Week 2: Perceived decrease in medication | One assessment after 2nd week of use
  Week 2: To assess whether use of RHINIX has led to a perceived decrease in use of medication.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Sigsgaard, Prof MD, Principal Investigator — Aarhus University, School of Public Health, Dept. of Environmental & Occupational Medicine
Locations (1):
- Aarhus University, School of Public Health, Department of Environmental & Occupational Medicine, Aarhus, Denmark

REFERENCES:
- [Derived] Kenney P, Hilberg O, Sigsgaard T. Clinical Application of Nasal Filters: An Observational Study on the Usability of Nasal Filters in Managing Seasonal Allergic Rhinitis. J Allergy Clin Immunol Pract. 2016 May-Jun;4(3):445-452.e4. doi: 10.1016/j.jaip.2016.01.003. Epub 2016 Feb 18. PMID 26897304